CLINICAL TRIAL: NCT06680037
Title: A Phase 1, Open-label Study to Evaluate the Safety and Clinical Activity of Azercabtagene Zapreleucel in Participants With B-cell Mediated Autoimmune Disorders
Brief Title: A Study to Assess the Safety and Clinical Activity of Azer-cel in Participants With B-cell Mediated Autoimmune Disorders
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TG-Azercel-101
Record Dates: First submitted 2024-11-01; First posted 2024-11-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: B-cell Mediated Autoimmune Disorders
Keywords: Progressive forms of multiple sclerosis (PMS); Primary Progressive MS (PPMS); Secondary Progressive MS (SPMS); Multiple Sclerosis (MS); Neuromyelitis optica spectrum disorder (MNOSD); Myasthenia Gravis (MG); Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Myasthenia Gravis; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azer-cel (Experimental): Participants will receive single dose of intravenous (IV) infusion of azer-cel at different dose levels, on Day 0 of the treatment period.
  Interventions: Drug: Azercabtagene zapreleucel (azer-cel)

INTERVENTIONS:
Drug: Azercabtagene zapreleucel (azer-cel) — IV infusion

SUMMARY:
The main objective of the study is to determine the recommended phase 2 dose (RP2D) of Azercabtagene zapreleucel (azer-cel).

ELIGIBILITY:
Inclusion Criteria:

1. Participants with Progressive forms of Multiple Sclerosis including Primary Progressive and Secondary Progressive MS.
2. Participants must have discontinued disease modifying therapy (DMT) prior to signing the ICF and meet the following washout criteria prior to receiving lymphodepletion.

Exclusion Criteria:

1. History of malignancy that has not been in remission for at least 2 years.
2. Viral Screening

   1. Evidence of chronic active or history of hepatitis B virus (HBV).
   2. Seropositive for human immunodeficiency virus (HIV) antibody.
3. History of bone marrow/hematopoietic stem cell or solid organ transplantation.
4. Prior treatment with adoptive T-cell therapy or any gene therapy product directed at any target (e.g. CAR T-cell therapy).

Note: Other protocol-specified Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLTs) | From Day 0 to Day 28
  DLT will be determined using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs), Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) | Up to Day 720
Change From Baseline in CAR T-cell Toxicities | Baseline, up to Day 720
Pharmacokinetics (PK) Plasma Concentrations of Azer-cel | Up to Day 720
Pharmacodynamics (PD) Plasma Concentrations of Azer-cel | Up to Day 720
Time to Confirmed Disability Progression (CDP) | Up to Day 720
Time to Confirmed Disability Improvement (CDI) | Up to Day 720
Change From Baseline in Brain MRI Gadolinium Enhancing T1, New or Enlarging Hyperintense T2 | Baseline, up to Day 720
Change From Baseline in Whole Brain Atrophy | Baseline, up to Day 720
Change From Baseline in Modified Rankin Scale (mRS) | Baseline, up to Day 720
Change From Baseline in Visual Acuity on Landolt C Broken Ring Chart (Low Contrast Visual Acuity [LCVA]) and High Contrast Visual Acuity (HCVA) | Baseline, up to Day 720
Change from Baseline in Myasthenia Gravis Activities of Daily Living Profile (MG-ADL) Total Score | Baseline, up to Day 720
Change from Baseline in the Revised 15-Component Myasthenia Gravis Quality of Life (MG-QOL15r) | Baseline, up to Day 720
Time to Relapse, as Defined by a 1 Point Change in Adjusted Inflammatory Neuropathy Cause and Treatment (aINCAT) | Baseline, up to Day 720
Change From Baseline in Inflammatory Neuropathy Cause and Treatment (INCAT) Score | Baseline, up to Day 720

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - TG Therapeutics Investigational Trial Site, La Jolla, California
  - TG Therapeutics Investigational Trial Site, Lexington, Kentucky
  - TG Therapeutics Investigational Trial Site, Ann Arbor, Michigan
  - TG Therapeutics Investigational Trial Site, Omaha, Nebraska
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial Site, Cleveland, Ohio
  - TG Therapeutics Investigational Trial Site, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No